**Official Title:** A Phase 3 Multicenter, Single-Arm, Open-Label Study Evaluating the Safety, Tolerability and Efficacy of StrataGraft® Construct in Pediatric Subjects with Deep Partial Thickness (DPT) Thermal Burns

NCT Number: NCT05517902

Document, Version and Date: Statistical Analysis Plan, Version 1.0, 03 July 2024



9201 Corporate Boulevard Suite 350

Rockville, MD 20850

Tel.: (301)294-6226 Fax: (301)294-4561

Email:

## Memo

| То: | Trial Master File – 01 DIA eTMF_Gen Section Statistical Analysis Plan | on - 11 Statistics - 11.01 Statistics Oversight - 11.01.01 |
|---|---|---|
| From: | | |
| CC: | | |
| Date: | 03Jul2024 | |
| Re: <i>M</i> | NK15011001 – Statistical Analysis Plan | 10 |

As of January 2024, the decision was made to close enrollment to the MNK15011001 study. Due to only 1 subject enrolled in the study, there will be no formal analyses performed on the study data. As such, this memo serves as the Statistical Analysis Plan (SAP).

Listings will be produced for all data collected from the eCRF and external laboratory transfers for subject subject. No other outputs are planned.

A table of contents of the planned output is in the following table. The file name will be provided as the [text].pdf with corresponding program file [text].txt. Study Data Tabulation Model (SDTM) datasets will be provided as .sas7bdat and .xpt files with corresponding specifications as an Excel file. Per the sponsor, there will be no ADaM datasets, define.xml files, reviewer's guides, nor SDTM annotated eCRF required. All datasets, planned output, and corresponding SAS programs will be provided to the sponsor via Mallinckrodt Secure File Transfer Protocol (SFTP) and will not be filed in the eTMF.

## Planned Output:

| Number | Title | CRFs / Data Source | File Name (.pdf) and |
|---|---|---|---|
| | | | Program Name (.txt) |
| Listing 16.2.1 | Screening Status | Screen Status | I-16-2-1-screen |
| <b>Listing 16.2.2</b> | <b>Protocol Deviations</b> | Protocol Deviations, | I-16-2-2-dv |
| | | Protocol Deviation Clinical | |
| | | Trial Management System | |
| | | (CTMS) Transfer | |

DP Clinical, Inc.


043Jul2024 

| Number | Title | CRFs / Data Source | File Name (.pdf) and<br>Program Name (.txt) |
|---|---|---|---|
| Listing 16.2.3.1 | Subject Disposition | Informed Consent,<br>Enrollment, Protocol<br>Reconsent, End of Study | I-16-2-3-1-ds |
| Listing 16.2.3.2 | Date of Visit | Date of Visit, Continuing to Visit | I-16-2-3-2-visit |
| Listing 16.2.3.3 | Log Summary | Log Summary | I-16-2-3-3-log |
| Listing 16.2.4.1 | Demographics | Demographics, Child<br>Bearing Potential | l-16-2-4-1-dm |
| Listing 16.2.4.2 | Medical History | Medical History | I-16-2-4-2-mh |
| Listing 16.2.4.3.1 | Prior and<br>Concomitant<br>Medications | Concomitant Medications | I-16-2-4-3-1-cm |
| Listing 16.2.4.3.2 | Concomitant<br>Procedures | Concomitant Procedures | I-16-2-4-3-2-cp |
| Listing 16.2.4.3.3 | Non-Drug<br>Therapies | Non-Drug Therapies | I-16-2-4-3-3-non-<br>drug |
| Listing 16.2.4.4 | Acute Burn History | Acute Burn History | l-16-2-4-4-bh |
| Listing 16.2.4.5 | Burn Wounds at<br>Screening and Re-<br>Assessment | Burn Wounds at<br>Screening, Re-Assessment<br>of Burn Wounds | l-16-2-4-5-bw |
| Listing 16.2.4.6 | Study Treatment<br>Site Identification | Study Treatment Site<br>Identification | l-16-2-4-6-trt-id |
| Listing 16.2.4.7 | Photography of<br>Study Treatment<br>Sites | Photography of Study<br>Treatment Sites | I-16-2-4-7-photo |
| Listing 16.2.5.1 | Treatments for<br>Other Non-Study<br>Site Burn Areas | Treatments for Other<br>Non-Study Site Burn<br>Areas | I-16-2-5-1-trt-other |
| Listing 16.2.5.2 | Study Treatment<br>Placement | Study Treatment<br>Placement | I-16-2-5-2-trt-place |
| Listing 16.2.5.3 | StrataGraft Disposition | StrataGraft Disposition | I-16-2-5-3-strata-disp |
| Listing 16.2.5.4 | StrataGraft Thaw<br>Time and Supply | StrataGraft Thaw Time and Supply | I-16-2-5-4-strata-<br>thaw |
| Listing 16.2.5.5 | Solutions Used | Solutions Used | I-16-2-5-5-solution |
| Listing 16.2.5.6 | Additional Autografting of Treatment Sites | Additional Autografting of<br>Treatment Sites | I-16-2-5-6-add-auto |
| Listing 16.2.6.1 | Infection<br>Assessment of | Infection Assessment of<br>Study Treatment Sites | l-16-2-6-1-inf |

DP Clinical, Inc.  03Jul2024 

| Number | Title | CRFs / Data Source | File Name (.pdf) and<br>Program Name (.txt) |
|---|---|---|---|
| | Study Treatment<br>Sites | | |
| Listing 16.2.6.2 | Wound Closure<br>Assessment | Wound Closure,<br>Continued Wound Closure<br>Assessment | I-16-2-6-2-wc |
| Listing 16.2.6.3.1 | Initial Study Site<br>Hospitalization | Initial Study Site<br>Hospitalization | I-16-2-6-3-1-init-hosp |
| Listing 16.2.6.3.2 | Additional<br>Hospitalizations | Additional<br>Hospitalizations | l-16-2-6-3-2-add-<br>hosp |
| Listing 16.2.6.4 | POSAS – Patient<br>Scale | POSAS – Patient Scale | l-16-2-6-4-posas |
| Listing 16.2.6.5 | POSAS – Observer<br>Scare Assessment<br>Questionnaire | POSAS – Observer Scare<br>Assessment<br>Questionnaire | l-16-2-6-5-posas |
| Listing 16.2.6.6 | PSAQ – Patient Scar<br>Assessment<br>Questionnaire | PSAQ – Patient Scar<br>Assessment<br>Questionnaire | I-16-2-6-6-psaq |
| Listing 16.2.6.7 | Evendol Pain Scale | Evendol Pain Scale | I-16-2-6-7-evandol |
| Listing 16.2.6.8 | Pain Assessment | Pain Assessment | I-16-2-6-8-pain |
| Listing 16.2.7.1 | Adverse Events | Adverse Events | I-16-2-7-1-ae |
| Listing 16.2.7.2 | Serious Adverse<br>Events | Adverse Events | I-16-2-7-2-sae |
| Listing 16.2.7.3 | Adverse Events Leading to Discontinuation | Adverse Events | I-16-2-7-3-aedisc |
| Listing 16.2.8.1 | Chemistry<br>Laboratory Results | Lab Summary, Local<br>Chemistry, Lab Vendor<br>Transfer | l-16-2-8-1-chem |
| Listing 16.2.8.2 | Hematology<br>Laboratory Results | Lab Summary, Local<br>Hematology, Lab Vendor<br>Transfer | l-16-2-8-2-hema |
| Listing 16.2.8.3 | Immunogenicity Laboratory Results | Lab Summary, Lab Vendor<br>Transfer | l-16-2-8-3-immu |
| Listing 16.2.8.4 | Archival Sample<br>Collection | Archival Sample<br>Collection | I-16-2-8-4-arch |
| Listing 16.2.8.5 | Pregnancy Test | Pregnancy Test | I-16-2-8-5-preg |
| <b>Listing 16.2.9</b> | Vital Signs | Vital Signs | I-16-2-9-vs |
| Listing 16.2.10 | Physical Examination | Physical Examination | l-16-2-10-pe |

DP Clinical, Inc.  03Jul2024 

| Signatures: | | | |
|---|---|---|---|
| DocuSigned by: Signer Name: Signing Reason: Tapprove this document Signing Time: 03-Jul-2024 2:14:30 PM EDT AB5E0253680E41C5AC79F08422C0D 1AF | | | 03-Ju1-2024 |
| | | Date: | 03-Ju1-2024 |
| , MS<br>DP Clinical, Inc. | | Date. | |
| DocuSigned by: Signer Name: Signing Reason: I approve this document Signing Time: 03-Jul-2024 2:58:24 PM EDT | | 10) | |
| 9CCE0059152345B2922510379343B57D | | Date: | 03-Ju1-2024 |
| , MPH<br>DP Clinical, Inc. | | | |
| | A. | | |
| DocuSigned by: Signer Name: Signing Reason: Iapprove this document Signing Time: 03-Jul-2024 2:23:59 PM EDT 98C58F586F5840ADBEC537D88147FC1B | Y | | |
| 9 | | Date: | 03-Ju1-2024 |
| DD CI: : I I | | | |
| DP Clinical, Inc. | | | |

DP Clinical, Inc. 

Downloaded by

## Sponsor:



03-Ju1-2024 Date:

, PhD

**Mallinckrodt Pharmaceuticals** 



DP Clinical, Inc. 